CLINICAL TRIAL: NCT01852279
Title: Brain Computer Interface Control of Functional Electrical Stimulation for a Hand Therapy in Tetraplegic Patients
Brief Title: BCI and FES for Hand Therapy in Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GN12NE574
Record Dates: First submitted 2013-04-30; First posted 2013-05-13 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active muscle stimulation (Experimental): Muscle stimulation delivered by Brain Computer Interface
  Interventions: Device: BCI-FES
- Passive muscle stimulation (Active Comparator): FES will be delivered by therapist
  Interventions: Device: Passive muscle stimulation

INTERVENTIONS:
Device: BCI-FES — Brain computer Interface delivered Function Electrical Stimulation
  Arms: Active muscle stimulation
Device: Passive muscle stimulation — Functional Electrical stimulation delivered by therapist
  Arms: Passive muscle stimulation

SUMMARY:
This study will assess whether functional recovery of the hand muscles in patients with spinal cord injury is enhanced when electrical stimulation of the muscles is delivered actively by means of using the electroencephalography wave patterns arising from the patient imagining moving their hand to operate the stimulator. A control group will obtain the electrical stimulation treatment passively by a therapist operating the machine.

DETAILED DESCRIPTION:
Injuries of the higher levels of the spinal cord, called tetraplegia, result in a complete or partial paralysis of both legs and arms, making the person dependent on their caregivers for elementary activities of daily living (ADL) such as drinking and feeding. About 60% of tetraplegics have an incomplete injury and can partially recover their movement and sensation. The success of a recovery greatly depends on the therapy within the first year after the injury. Functional electrical stimulation (FES) is a relatively novel therapy of the hand. In FES therapy electrodes are attached on the surface the patients's forearms and electrical current is delivered through them. A disadvantage of the current FES therapy is that a therapist has to switch the stimulator on and off because patients cannot use either of their hands. In our previous pilot study performed on two acute tetraplegic patients we tested feasibility of using brain-computer interface (BCI) to control FES on patient's will. BCI is based on recording the patient's brain activity. BCI can detect the patient's intention to move the hand even if they are not able to physically move it. Using BCI, patients control the FES by thinking to move their hand.

A BCI-FES therapy will provide a simultaneous training of neural pathways from the brain to the hand muscle (motor imagination/attempt) and from the muscle to the brain (electrical stimulation of muscles). This form of therapy could promote faster and more complete recovery

In this controlled study we aim to provide a BCI-FES therapy to both chronic and subacute tetraplegic patients over a period of 20 sessions and to access the functional and neurological outcome of the therapy. Five chronic patients (more than a year after the injury) will participate in a cross-over study as we do not expect that they will recover spontaneously without BCI-FES. Subacute patients will be receiving both a conventional therapy and BCI-FES so recovery can be caused by either of these two therapies. Therefore it is necessary to have a treatment and a control group. Each group will have 10 patients, age and injury matched. Both groups will receive the same amount of electrical stimulation but only the treatment group will voluntarily control the electrical stimulator using BCI. A control group will receive passive electrical stimulation of the same hand muscles but without using BCI.

ELIGIBILITY:
Inclusion Criteria:

* incomplete (ASIA B, C) tetraplegia with injury at level C4-C8
* aged between 18 and 70 years old
* a candidate suitable for the conventional therapy

Exclusion Criteria:

* Patients must not have presence of any neurological problem that might distort recording standard brain signal during motor imagination (example: brain damage, epilepsy, Parkinson disease and multiple sclerosis)
* Patients must not have cognitive impairments (hearing, vision and general inability to understand instructions)
* Patients must not suffer from recurring pressure sore which prevent patient from sitting for at least an hour
* Patients must not suffer from excessive spasm that would increase with electrical stimulation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-05-08 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Muscle strength as measured by the Oxford manual test | Between initial and final assessment after up to 8 weeks of treatment

SECONDARY OUTCOMES:
Changes in patients EEG before and after each treatment session | between beginning and end of each one hour treatment session
  Measures will be taken at the beginning and end of each of the 20 treatment sessions
Difference in EEG between the treatment and the control group | Between initial and final assessment after up to 8 weeks of treatment
Difference in Somatosensory evoked potential between the treatment and control group | Between initial and final assessment after up to 8 weeks of treatment
Difference in somatosensory evoked potential before and after a treatment session | Between initial and final assessment after up to 8 weeks of treatment
Patient's experience of using BCI-FES | Between initial and final assessment after up to 8 weeks of treatment
  A questionnaire will collect information
Quadriplegia index of function | Between initial and final assessment after up to 8 weeks of treatment
Range of movement of wrists and fingers | Between initial and final assessment after up to 8 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Vuckovic, PhD, Principal Investigator — University of Glasgow
Locations (1):
- Queen Elizabeth National Spinal Injuries Unit, Glasgow, United Kingdom

REFERENCES:
- [Derived] Osuagwu BC, Wallace L, Fraser M, Vuckovic A. Rehabilitation of hand in subacute tetraplegic patients based on brain computer interface and functional electrical stimulation: a randomised pilot study. J Neural Eng. 2016 Dec;13(6):065002. doi: 10.1088/1741-2560/13/6/065002. Epub 2016 Oct 14. PMID 27739405